CLINICAL TRIAL: NCT01911585
Title: Efficacy of 60-minute Versus 90-minute Sessions in Treating PTSD Using Prolonged Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 817717
Record Dates: First submitted 2013-07-22; First posted 2013-07-30 (Estimated); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Posttraumatic Stress Disorder; PTSD
Keywords: Posttraumatic Stress Disorder; PTSD; Prolonged Exposure Therapy; Cognitive Behavioral Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 90 minute Prolonged Exposure Sessions (Active Comparator): Prolonged Exposure Therapy for PTSD consists of 10 to 15 weekly or twice-weekly sessions, each lasting about 90 minutes, with 40 to 60 minutes imaginal exposure.
  Interventions: Behavioral: Prolonged Exposure Therapy
- 60 minute Prolonged Exposure Sessions (Experimental): This treatment condition is a modified version of Prolonged Exposure therapy for PTSD. It consists of 10 to 15 weekly or twice-weekly sessions, each lasting about 60 minutes, with 20 minutes imaginal exposure.
  Interventions: Behavioral: Prolonged Exposure Therapy

INTERVENTIONS:
Behavioral: Prolonged Exposure Therapy — Prolonged exposure therapy (PE), a specific exposure therapy program for PTSD is a highly effective treatment for PTSD. The key components of PE are imaginal exposure to the traumatic event and processing it (revisiting of the traumatic memory in imagination) followed by processing of the revisiting experience, and in vivo exposure to avoided trauma-related situations and objects.

SUMMARY:
The purpose of this study is to determine whether 60-minute sessions of prolonged exposure (PE) are as effective as the standard 90-minute session for treating posttraumatic stress disorder (PTSD). Participants will include patients ages 18 or older with a current diagnosis of PTSD who are seeking treatment in our clinic. Patients who have current substance dependence, psychosis, and suicidal ideation with intent and plan may not be suitable for receiving PE and may be offered another treatment or referred to a different treatment center. Participants will be randomized to receive either the 90- minute or 60-minute PE session. A blind evaluator will assess for pre-treatment, post-treatment, and follow-up levels of symptom severity using the PTSD Symptoms Scale Interview (PSS-I). Participants will attend weekly treatment sessions with any of our faculty members and will complete self-report measures at every session (see below).

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of PTSD
* Recommended by therapist to receive Prolonged Exposure therapy

Exclusion Criteria:

* Current substance dependence, psychosis, suicidal ideation with intent and plan, or other psychiatric problems warranting immediate clinical attention or would interfere with Prolonged Exposure therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in PTSD Symptom Scale, Interview Version (PSS-I; Foa, Riggs, Dancu, & Rothbaum, 1993; Powers, Gillihan, Rosenfield, Jerud & Foa, 2012) | Pre-treatment through 6 month follow-up
  The PSS-I will be administered on 4 separate occasions We will measure the change in PSS-I scores from pre-treatment to post-treatment, 3 month follow-up, and 6 month follow-up.
  The PSS-I is a 20-minute, 17-item clinical interview that evaluates DSM-IV PTSD symptoms on a frequency/severity scale. The interview yields a full-scale score and subscales for each of the three PTSD symptom clusters. Psychometric studies revealed internal reliability of .91 for the full scale, and .78, .80, and .82 for the reexperiencing, avoidance and arousal clusters (Foa & Tolin, 2000).

SECONDARY OUTCOMES:
Posttraumatic Diagnostic Scale (PDS; Foa et al., 1997) | Pre-treatment through 6 months post-treatment
  The PDS will be administered at every other treatment session and at post-treatment, 3 month follow-up, and 6 month follow-up. The measure will be used to closely monitor treatment progress and help assess severity of symptoms.
  The PDS is a 17-item self-report measure that provides total and subscale severity scores and categorical classification of PTSD. The PDS demonstrated high internal consistency (.92 total, .78 re-experiencing, .84 avoidance, and .84 hyperarousal). Test-retest reliability is good, ranging from .74 to .85. High diagnostic agreement (82%) with the SCID-IV was noted: sensitivity was .89, and specificity, .75. The PDS is highly related to other measures of trauma related psychopathology. Participants will complete this measure at the beginning of every other treatment session.
Beck Depression Inventory (BDI; Beck et al., 1961) | Pre-treatment through 6 month follow-up
  The BDI will be administered at every other treatment session and at post-treatment, 3 month follow-up, and 6 month follow-up. The measure will be used to closely monitor treatment progress and help assess severity of symptoms.
  The BDI is a 21-item scale assessing depression. The inventory's internal consistency ranges from .58 to .93, test-retest reliability ranges from .69 to .90. Participants will complete this report measure at the beginning every other treatment session.
Post-Traumatic Cognitions Inventory (PTCI; Foa et al., 1999) | Pre-treatment through 6 month follow-up
  The PTCI will be administered at every other treatment session and at post-treatment, 3 month follow-up, and 6 month follow-up. The measure will be used to closely monitor treatment progress and help assess severity of symptoms.
  This 36-item instrument assesses post-trauma cognitions across self, world, and self-blame and yields a total score. The scale has high internal consistency (.97, .88, .86, 97, respectively) and correlates well with PTSD severity, anxiety, and depression (.44 to .79). This 36-item instrument assesses dysfunctional post trauma cognitions theoretically thought to underlie the development of PTSD. Participants will complete this measure at the beginning of every treatment session.

CONTACTS AND LOCATIONS:
Overall Officials: Edna B. Foa, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Center for the Treatment and Study of Anxiety, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Foa EB, Bredemeier K, Acierno R, Rosenfield D, Muzzy W, Tuerk PW, Zandberg LJ, Hart S, Young-McCaughan S, Peterson AL, McLean CP. The efficacy of 90-min versus 60-min sessions of prolonged exposure for PTSD: A randomized controlled trial in active-duty military personnel. J Consult Clin Psychol. 2022 Jun;90(6):503-512. doi: 10.1037/ccp0000739. PMID 35771512